CLINICAL TRIAL: NCT02163954
Title: Platelet Reactivity in Patients With End Stage Renal Disease Receiving Clopidogrel Compared With Ticagrelor
Brief Title: ONSET and OFFSET of Ticagrelor in ESRD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyunghee University (Other)
Responsible Party: Principal Investigator, Weon Kim, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PIANO3; Seoul, Korea (Other Grant/Funding Number: 2010-0019913)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Kidney Disease
Keywords: platelet; ticagrelor; clopidogrel; end stage renal disease; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Active Comparator): Patients treated with clopidogrel for 14 days
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel
- Ticagrelor (Experimental): Patients treated with ticagrelor for 14 days
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — After randomization, an initial loading dose of ticagrelor (180 mg) was given and maintenance doses (ticagrelor 90 mg twice daily) was treated for 14 days.
  Other Names: Ticagrelor (Brilinta)
Drug: Clopidogrel — After randomization, an initial loading dose of clopidogrel (300 mg) was given and maintenance doses (clopidogrel 75 mg once daily) was treated for 14 days.
  Other Names: Clopidogrel (Plavix)

SUMMARY:
Patients with severe chronic kidney disease or end stage renal disease (ESRD) on hemodialysis (HD) exhibited higher platelet reactivity to clopidogrel than did those with normal renal function. Not enough study has been conducted about the antiplatelet effects of ticagrelor in these cardiovascular high risk patients. We hypothesized ticagrelor would achieve more and faster antiplatelet effects compared with clopidogrel in ESRD patients on HD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a strong risk factor for cardiovascular morbidity and mortality, and confers an increasing risk of stent thrombosis even when dual antiplatelet therapy (clopidogrel and aspirin) is administered. Recently, we demonstrated that patients with severe CKD or end stage renal disease (ESRD) on hemodialysis (HD) exhibited higher platelet reactivity to clopidogrel than did those with normal renal function. One of good option to overcome high platelet reactivity in ESRD patients would be ticagrelor which has been already shown improved clinical outcomes. But little is known the antiplatelet effects of ticagrelor in ESRD patients on HD. The present study was designed to determine the antiplatelet effect as well as the onset and offset action of ticagrelor compared with clopidogrel in patients with ESRD undergoing maintenance HD.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients undergoing regular (≥ 6 months) maintenance HD
* ongoing (≥ 2 months) treatment with clopidogrel
* P2Y12 reaction units (PRUs) were more than 235

Exclusion Criteria:

* known allergies to aspirin, clopidogrel, or ticagrelor
* concomitant use of other antithrombotic drugs (oral anticoagulants, dipyridamole)
* thrombocytopenia (platelet count <100,000/mm3)
* hematocrit <25%
* uncontrolled hyperglycemia (hemoglobin A1c >10%)
* liver disease (bilirubin level >2 mg/dl)
* symptomatic severe pulmonary disease
* active bleeding or bleeding diathesis
* gastrointestinal bleeding within the last 6 months
* hemodynamic instability
* acute coronary or cerebrovascular event within the last 3 months
* pregnancy
* any malignancy
* concomitant use of a cytochrome P450 inhibitor or nonsteroidal anti-inflammatory drug
* recent treatment (<30 days) with a glycoprotein IIb/IIIa antagonist

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The difference of antiplatelet effects assessed by VerifyNow assay | 14 days after study drug treatment
  The difference of PRU values achieved following antiplatelet therapy

SECONDARY OUTCOMES:
the rate of onset and offset of the antiplatelet effects | 14 days after study drugs treatment
  the difference of slope during onset and offset of study drugs

OTHER OUTCOMES:
Adverse events | during study period
  Adverse events such as bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, MD, PhD, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730